CLINICAL TRIAL: NCT07332416
Title: Pilot Study of Continuous Glucose Monitoring for Postpartum Glucose Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medstar Health Research Institute (Other); University of North Carolina, Chapel Hill (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00143138; P30DK124723 (NIH)
Record Dates: First submitted 2026-01-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes
Keywords: Continuous glucose monitoring; Postpartum glucose screening; Dysglycemia
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Postpartum CGM (Active Comparator): Postpartum continuous glucose monitoring
  Interventions: Other: Continuous glucose monitoring for 14 days using the Freestyle LibrePro by Abbott
- Postpartum OGTT (No Intervention): Postpartum oral glucose tolerance test
- No screening (No Intervention): No postpartum glucose screening

INTERVENTIONS:
Other: Continuous glucose monitoring for 14 days using the Freestyle LibrePro by Abbott — Postpartum CGM
  Arms: Postpartum CGM

SUMMARY:
The oral glucose tolerance test (OGTT) is the standard of care in the postpartum period to screen patients with gestational diabetes mellitus (GDM) for persistent dysglycemia. However, most patients find it burdensome and dread having to do it. Adherence rates are low (18-61%), impeding initiation of follow-up care to improve diabetes-related outcomes in subsequent pregnancies and long-term.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) is an appealing alternative to the OGTT because it is a low-burden, fully remote, comprehensive assessment of glycemic status. Emerging data suggest that CGM is superior to the OGTT in identifying persistent dysglycemia at 2-5 months postpartum, and preferable to the OGTT among women willing to complete both assessments in the context of a research study. This study proposes a feasibility study of postpartum CGM among patients who do not complete the standard postpartum OGTT. The study will offer CGM in a telehealth (fully remote) context to determine if it can increase adherence to postpartum glycemic screening in real-world settings. This study will (a) evaluate uptake of CGM screening, (b) characterize patients who complete CGM, complete the OGTT, or do not complete screening, and (c) monitor initiation of follow-up care after abnormal results.

ELIGIBILITY:
Inclusion Criteria:

* 12-16 weeks postpartum
* Gestational diabetes Mellitus (GDM) diagnosis in most recent pregnancy
* Oral Glucose Tolerance Test (OGTT) order placed in the medical record

Exclusion Criteria:

* Pre-gestational diabetes
* Non-English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postpartum
Enrollment: 1300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Continuous Glucose Monitor (CGM) uptake - Percentage of CGM-eligible patients | 20 weeks postpartum
  Percentage of CGM-eligible patients that return a used CGM sensor

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Sauder, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be published from this pilot study; individual patient level data will be kept confidential.